CLINICAL TRIAL: NCT02043275
Title: Effect of a Resistance Training Program on the Jump Landing Biomechanics of Young Female Athletes
Brief Title: Effect of Resistance Training on Jump Landing Mechanics in Young Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joanne Parsons, PhD Candidate, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #E2013:015; CIHR (Other Grant/Funding Number: Application #:237137)
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: resistance training
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leg training (Experimental): Lower body resistance training only
  Interventions: Other: Leg training
- Arm training (Active Comparator): Upper body resistance training only
  Interventions: Other: Arm training

INTERVENTIONS:
Other: Leg training — Lower body resistance training twice per week for one hour each time.
  Arms: Leg training
Other: Arm training — Upper body resistance training twice per week for one hour each time.
  Arms: Arm training

SUMMARY:
The purpose of this study is to determine if jump landing mechanics in young female athletes can be improved with a resistance training intervention.

DETAILED DESCRIPTION:
After initial baseline testing, athletes were randomly selected to receive upper body (control group) or lower body (intervention group) resistance training. Athletes attended supervised training sessions twice per week for 12 weeks, after which they were re-tested.

ELIGIBILITY:
Inclusion Criteria:

* at least one year experience playing organized sports

Exclusion Criteria:

* previous experience with resistance training
* any injury with a pain level of more than 3/10 on VAS
* any health condition that would preclude them from completing the training or testing
* previous experience using a Biodex dynamometer

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Landing Error Scoring System score from Baseline to 12 weeks. | Baseline and 12 weeks

SECONDARY OUTCOMES:
Neuromuscular power of the hip abductors measured by a Biodex isokinetic dynamometer | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Parsons, PhD Cand., Principal Investigator — University of Manitoba; Michelle M Porter, PhD, Study Director — University of Manitoba
Locations (1):
- Faculty of Kinesiology and Recreation Management, Winnipeg, Manitoba, Canada